CLINICAL TRIAL: NCT04087187
Title: A Randomized, 3-period, 3-treatment, Single-dose, Open-label, Single-center, Crossover Study to Assess the Pharmacokinetics of 3 Doses of AZD5718
Brief Title: A Study to Assess the Drug Absorption Into the Blood After Administration of 3 Doses of AZD5718
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7550C00009
Record Dates: First submitted 2019-08-19; First posted 2019-09-12 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
Keywords: Pharmacokinetics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The following treatments will be given in crossover design:
  * Treatment A: AZD5718 Dose A tablet
  * Treatment B: AZD5718 Dose B tablet
  * Treatment C: AZD5718 Dose C tablet
  There will be 6 arms consisting of all possible treatment sequences. The treatment sequence per arm will be:
  Arm1: ABC Arm2: ACB Arm3: BAC Arm4: BCA Arm5: CAB Arm6: CBA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm1: AZD5718 Dose A + AZD5718 Dose B + AZD5718 Dose C (Experimental): Subjects will receive one tablet once daily (QD) of each treatment according to treatment arm.
  Treatment A: AZD5718 Dose A, Treatment B: AZD5718 Dose B, Treatment C: AZD5718 Dose C, with a minimum washout period of 4 days between each dose administration.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Arm2: AZD5718 Dose A + AZD5718 Dose C + AZD5718 Dose B (Experimental): Subjects will receive one tablet once daily (QD) of each treatment according to treatment arm.
  Treatment A: AZD5718 Dose A, Treatment C: AZD5718 Dose C, Treatment B: AZD5718 Dose B, with a minimum washout period of 4 days between each dose administration.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Arm3: AZD5718 Dose B + AZD5718 Dose A + AZD5718 Dose C (Experimental): Subjects will receive one tablet once daily (QD) of each treatment according to treatment arm.
  Treatment B: AZD5718 Dose B, Treatment A: AZD5718 Dose A, Treatment C: AZD5718 Dose C, with a minimum washout period of 4 days between each dose administration.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Arm4: AZD5718 Dose B + AZD5718 Dose C + AZD5718 Dose A (Experimental): Subjects will receive one tablet once daily (QD) of each treatment according to treatment arm.
  Treatment B: AZD5718 Dose B, Treatment C: AZD5718 Dose C, Treatment A: AZD5718 Dose A, with a minimum washout period of 4 days between each dose administration.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Arm5: AZD5718 Dose C + AZD5718 Dose A + AZD5718 Dose B (Experimental): Subjects will receive one tablet once daily (QD) of each treatment according to treatment arm.
  Treatment C: AZD5718 Dose C, Treatment A: AZD5718 Dose A, Treatment B: AZD5718 Dose B, with a minimum washout period of 4 days between each dose administration.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Arm6: AZD5718 Dose C + AZD5718 Dose B + AZD5718 Dose A (Experimental): Subjects will receive one tablet once daily (QD) of each treatment according to treatment arm.
  Treatment C: AZD5718 Dose C, Treatment B: AZD5718 Dose B, Treatment A: AZD5718 Dose A, with a minimum washout period of 4 days between each dose administration.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — Subject will be given AZD5718 Dose A tablet once daily
Drug: Treatment B — Subjects will be given AZD5718 Dose B tablet once daily
Drug: Treatment C — Subjects will be given AZD5718 Dose C tablet once daily

SUMMARY:
This study will be conducted to evaluate the AZD5718 pharmacokinetic (PK) doses in order to determine exposure in a new dose range and compare with previous results. This study will include 14 subjects in a single site in United Kingdom. Each subject will be involved in the study for 6 to 7 weeks.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, 3-period, 3-treatment, crossover study performed in healthy subjects at a single study center.

A total of 14 healthy male and female subjects (of no childbearing potential) will be randomized to ensure that at least 12 subjects are evaluable. Each subject will receive 3 different treatments at least 4 days apart and will be dosed following an overnight fast of at least 10 hours. The following treatments will be given:

* Treatment A: AZD5718 Dose A tablet
* Treatment B: AZD5718 Dose B tablet
* Treatment C: AZD5718 Dose C tablet

The study will comprise:

* A Screening Period of maximum 28 days.
* Three Treatment Periods during which subjects will be resident from the day before first dosing with AZD5718 (Day -1) in Treatment Period 1 until at least 48 hours after last dosing with AZD5718 in Treatment Period 3 for collection of PK and safety samples. Subjects will be discharged on Day 3 of Treatment Period 3.
* A Follow up Visit, 5 to 7 days after the last dose of investigational medicinal product (IMP).

There will be a minimum washout period of 4 days between each dose administration.

Each subject will be involved in the study for 6 to 7 weeks. This study will be conducted in male and female subjects aged 18 to 55 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and/or female subjects aged 18 to 55 years (inclusive at Screening Visit) with suitable veins for cannulation or repeated venipuncture.
* Males must be willing to use appropriate contraception methods.
* Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit (Day -1) must not be lactating and must be of non-childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria

  * Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the postmenopausal range.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
  * Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results at the Screening Visit and/or admission to the Clinical Unit (Day -1), as judged by the Investigator including:

  * Alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) >1.5 x ULN.
  * Bilirubin (total) >1.5 x ULN.
  * Gamma glutamyl transpeptidase (GGT) >1.5 x ULN.
* Any clinically significant abnormal findings in vital signs at the Screening Visit and/or admission to the Clinical Unit (Day -1), as judged by the Investigator.
* Any clinically significant abnormalities on 12 lead ECG at the Screening Visit, as judged by the Investigator.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Known or suspected history of drug abuse, as judged by the Investigator.
* Known or suspected Gilbert's syndrome.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the 3 administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.
* Plasma donation within 1 month of the Screening Visit or any blood donation/loss more than 500 mL during the 3 months prior to the Screening Visit.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to the Screening Visit.
* Excessive intake of caffeine containing drinks or food (eg, coffee, tea, chocolate,) as judged by the Investigator.
* Positive screen for drugs of abuse, alcohol or cotinine at the Screening Visit or on admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
* Subjects who have previously received AZD5718.
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Area under plasma concentration time curve from zero to infinity (AUC) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718
Pharmacokinetic parameter: Area under the plasma concentration curve from time zero to time of last quantifiable concentration (AUClast) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718
Pharmacokinetic parameter: Maximum observed plasma concentration (Cmax) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718
Pharmacokinetic parameter: Drug concentration 24 hours after dosing (C24) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718
Pharmacokinetic parameter: Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t1/2λz) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718
Pharmacokinetic parameter: Time to reach maximum observed plasma concentration (tmax) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718
Pharmacokinetic parameter: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To evaluate the pharmacokinetics and exposure of 3 different doses of AZD5718

SECONDARY OUTCOMES:
Number of subjects with advers event | Upto 7 weeks
  Number of subjects with adverse event and/or abnormal vital signs or physical examination or laboratory assessments to further assess the safety of single doses of AZD5718 in healthy subjects.
Pharmacokinetic parameter: AUC | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To assess dose proportionality of AZD5718
Pharmacokinetic parameter: Cmax | Day 1: Pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours post dose, Day 2: 24 and 36 hours post dose and Day 3: 48 hours post dose
  To assess dose proportionality of AZD5718

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom